CLINICAL TRIAL: NCT05807399
Title: A Multiple-arm, Multiple-stage (MAMS), Phase 2B/C, Open-label, Randomized, Controlled Platform Trial to Evaluate Experimental Arms Including Optimised Use of Existing and Introduction of Novel Anti-tuberculosis Drugs, in Adults With Newly Diagnosed, Drug-sensitive, Smear-positive Pulmonary Tuberculosis
Brief Title: PanACEA - STEP2C -01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Hoelscher (Other)
Collaborators: Radboud University Medical Center (Other); University of California, San Francisco (Other); University College, London (Other); GlaxoSmithKline (Industry); LigaChem Biosciences, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Michael Hoelscher, Prof. Dr., Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PanACEA - STEP2C -01
Record Dates: First submitted 2023-02-14; First posted 2023-04-11 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Tuberculosis; Other Specified Pulmonary Tuberculosis
Keywords: Tuberculosis, Pulmonary; Tuberculosis; Antitubercular Agents; Safety; Tolerability; Pharmacokinetics (PK); Moxifloxacin; BTZ-043; Rifampicin
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — 2-(2-methyl-1,4-dioxa-8-azaspiro(4.5)dec-8-yl)-8-nitro-6-(trifluoromethyl)-4H-1,3-benzothiazin-4-one; Rifampin; Isoniazid; Pyrazinamide; Moxifloxacin; GSK656; delpazolid; pretomanid; Ethambutol; Ethionamide

STUDY DESIGN:
Intervention Model Description: The study will compare the efficacy, safety of 5 experimental regimens with a standard control regimen in participants with newly diagnosed, drug sensitive pulmonary tuberculosis.
  In stage 1, participants will be randomly allocated to the control or one of the 2 rifampicin-containing experimental regimens in the ratio 1:1:1. In stage 2, the experimental arm 4 containing BTZ-043 will be added. The allocation ratio will be changed to co-enrol the remaining participants in arms 1- 3 simultaneously with arm 4 with an allocation ratio of 1:1:1:2. When arms 1-2 are fully enrolled and arm 4 is not, further participants will be randomized 1:1 to control and experimental arm 4. Not all countries will participate in stage 2.
  In stage 3, participants will be allocated in parallel to control arm treatment (now designated arm 7) or the experimental arms 5 and 6, favouring arm 5, 2:1:1 over arms 6 and control. This stage will start after completion of recruitment in the stages 1 and 2.
Who Masked: Outcomes Assessor
Masking Description: This study will be open-label, participants and physicians will be aware of treatment allocation. To ensure unbiased assessment of efficacy endpoints, the personnel assessing participants' outcomes, like the microbiology laboratory staff, will remain blinded to treatment assignment throughout the whole study. Every effort will be made to maintain this blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Arm 1 (Stage 1) (Experimental): Rifampicin 2100mg, isoniazid 300mg, pyrazinamide 1600mg moxifloxacin 600mg; given once daily for 17 weeks (R2100HZM600)
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Moxifloxacin
- Arm 2 (Stage 1) (Experimental): Rifampicin 2100mg, isoniazid 300mg, pyrazinamide 2000mg/2400mg, moxifloxacin 600mg; given once daily for 12 weeks (R2100HZoptM600)
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Moxifloxacin
- Arm 3 (Active Comparator): Stage 1: control arm (2HRZE-4RH) Stage 2: continuation of control-arm from STAGE 1 (2HRZE-4RH)
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Ethambutol (E)
- Arm 4 (Stage 2) (Experimental): Rifampicin, Isoniazid, and Pyrazinamide in weight-banded standard dosages with BTZ-043 1,000mg; given once daily for 17 weeks (RHZT), then rifampicin and isoniazid in weight-banded dosages; given once daily for 9 weeks (RH)
  Interventions: Drug: BTZ-043; Drug: Rifampicin; Drug: Isoniazid; Drug: Pyrazinamide
- Arm 5 (Stage 3) (Experimental): Alpibectir (GSK3729098) 45mg, ethionamide 500mg (A/Eto) with possibility of lower alpibectir and Eto doses based on emerging clinical data, from the ENABLE study [ Clinical Trials gov NCT06748937] and non-clinical data and endorsed by the GSK Global safety board, rifampicin, pyrazinamide and ethambutol at standard doses given once daily for 8 weeks, continued with RIF and INH at standard doses for 18 weeks.
  Interventions: Drug: Rifampicin; Drug: Pyrazinamide; Drug: Alpibectir (GSK3729098); Drug: Ethambutol (E); Drug: Ethionamide
- Arm 6 (Stage 3) (Experimental): Pretomanid 200mg, ganfeborole (GSK3036656) 20mg, BTZ-043 1000mg and delpazolid (LCB01-0371) 1200mg; given once daily for 26 weeks
  Interventions: Drug: BTZ-043; Drug: Ganfeborole (GSK3036656); Drug: Delpazolid (LCB01-0371); Drug: Pretomanid (Pa)
- Arm 7 (Stage 3) (Active Comparator): Parallel control arm (2HRZE-4RH)
  Interventions: Drug: Rifampicin; Drug: Isoniazid; Drug: Pyrazinamide; Drug: Ethambutol (E)

INTERVENTIONS:
Drug: BTZ-043 — BTZ-043 1000mg once daily in arms 4 and 6.
  Arms: Arm 4 (Stage 2); Arm 6 (Stage 3)
Drug: Rifampicin — Rifampicin will be dosed in a fixed high-dose (2100 mg for arms 1 and 2) or a weight-banded regular dose (10 mg/kg) in arm 3, 5 and 7.
  Arms: Arm 1 (Stage 1); Arm 2 (Stage 1); Arm 3; Arm 4 (Stage 2); Arm 5 (Stage 3); Arm 7 (Stage 3)
Drug: Isoniazid — Isoniazid will be dosed at fixed dose of 300mg in arms 1 and 2, and regular dose of 5 mg/kg in arm 3 and 7.
  Arms: Arm 1 (Stage 1); Arm 2 (Stage 1); Arm 3; Arm 4 (Stage 2); Arm 7 (Stage 3)
Drug: Pyrazinamide — Pyrazinamide will be dosed in a fixed regular dose in arm 1 (1600 mg), a weight banded high dose in arm 2 (2000/2400 mg) or a weight-banded regular dose (25 mg/kg) in arm 3, 5 and 7.
  Arms: Arm 1 (Stage 1); Arm 2 (Stage 1); Arm 3; Arm 4 (Stage 2); Arm 5 (Stage 3); Arm 7 (Stage 3)
Drug: Moxifloxacin — Moxifloxacin will be dosed at 600 mg orally once daily in arms 1-2.
  Arms: Arm 1 (Stage 1); Arm 2 (Stage 1)
Drug: Alpibectir (GSK3729098) — Alpibectir 45 mg OD plus Ethionamide 500 mg OD combined with rifampicin pyrazinamide and ethambutol at standard weight-banded doses in arm 5.
  Arms: Arm 5 (Stage 3)
Drug: Ganfeborole (GSK3036656) — Ganfeborole 20 mg OD in arm 6
  Arms: Arm 6 (Stage 3)
Drug: Delpazolid (LCB01-0371) — Delpazolid 1200mg OD in arm 6
  Arms: Arm 6 (Stage 3)
Drug: Pretomanid (Pa) — Pretomanid 20mg OD in arm 6.
  Arms: Arm 6 (Stage 3)
Drug: Ethambutol (E) — Ethambutol 20mg/Kg OD in arm 3, 5 and 7
  Arms: Arm 3; Arm 5 (Stage 3); Arm 7 (Stage 3)
Drug: Ethionamide — Ethionamide 500mg OD in arm 5.
  Arms: Arm 5 (Stage 3)

SUMMARY:
This is a phase 2B/C, open label platform study that will compare the efficacy, safety of experimental regimens with a standard control regimen in participants with newly diagnosed, drug sensitive pulmonary tuberculosis.

In stage 1, participants will be randomly allocated to the control or one of the 2 rifampicin-containing experimental regimens in the ratio 1:1:1.

In stage 2, the experimental arm 4 containing BTZ-043 will be added. The allocation ratio will be changed to co-enrol the remaining participants in arms 1- 3 simultaneously with arm 4 in a ratio of 1:1:1:2. When arms 1-2 are fully enrolled and arm 4 is not, further participants will be randomized 1:1 to control and experimental arm 4. Not all countries will participate in stage 2.

In stage 3, participants will be allocated in parallel to control arm treatment (now designated arm 7) or the experimental arms 5 and 6, favouring arm 5, 2:1:1 over arms 6 and control. This stage will start after completion of recruitment in the stages 1 and 2. Enrolment of participants into arm 5 will proceed following review of data from the ENABLE/UNITE-03 (NCT06748937), non-clinical safety data and after endorsement by the DSMB. Thus, arm 5 recruitment might start after arms 6 and 7, which may require an increase in the control arm sample size to ensure controls are recruited concomitantly.

DETAILED DESCRIPTION:
This open label, phase 2B/C , randomized, controlled platform trial, will evaluate experimental arms including regimens with optimized doses of rifampicin, pyrazinamide, and moxifloxacin; a regimen with BTZ-043 combined first-line anti-TB drugs; a regimen with alpibectir-boosted ethionamide replacing isoniazid in combination with first-line anti-TB durgs, and a bedaquiline sparing regimen containing new anti-TB drugs (ganfeborole, BTZ-043 and delpazolid) in adults with newly diagnosed, drug sensitive, smear-positive pulmonary tuberculosis

A total of up to 390 (270 for stage 1 and 2, and 120 for stage 3, respectively) adult (≥ 18 years of age) participants will be enrolled.

In case of a high number of dropouts or non-evaluable participants, it may be necessary to recruit more participants into the study.

Also, if the stage 2 starts later than stage 1, it may be necessary to increase the number of control arm participants to achieve a 1:1 ratio of concomitantly recruited control and arm 4 participants until the recruitment for arm 4 is completed (see sample size considerations).

Stage 3 will start after stages 1 and 2 complete recruitment.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written, informed consent prior to all trial-related procedures including HIV testing.
2. Male or female, aged between 18 and 65 years, inclusive.
3. Body weight (in light clothing and with no shoes) between 40 and 90 kg, inclusive.
4. Newly diagnosed, previously untreated, drug susceptible pulmonary TB: presence of MTB complex and rapid molecular tests result confirming susceptibility to RIF and INH such as GeneXpert and/or HAIN MTBDR plus. Participants who had a previous history of TB may be enrolled in this trial, if they:

   * had a good treatment response in the opinion of the investigator; i.e. TB symptoms improved sufficiently or resolved suggesting a cure of the past episode; AND
   * no persistent microbiological positivity is seen (in case microbiological results are available); AND - their treatment course was completed AND
   * the last dose of treatment was more than 3 months ago.
5. A chest X-ray (no older than 2 weeks) which shows abnormalities that, in the opinion of the Investigator, are consistent with TB.
6. Sputum positive on microscopy from concentrated sputum for acid-fast bacilli (at least 1+ on the IUATLD/WHO scale) AND/OR positive GeneXpert MTB/RIF Ultra® semi-quantitative result "medium" or "high" on at least one sputum sample.
7. The participant understands the interaction between the study drugs and certain foods and is willing to forgo the consumption of those foods for the period of study medication.
8. The participant is not of child-bearing potential or is willing to use effective methods of contraception when engaging in heterosexual intercourse, as defined below:

   1. Non-childbearing potential:

   i. Female participant/sexual partner of male participant: Bilateral oophorectomy, and/or hysterectomy or bilateral tubal ligation more than 12 months ago and/or has been postmenopausal with a history of no menses for at least 12 consecutive months and confirmed by a FSH test.

   ii. Male participant/sexual partner of female participant: Vasectomised or has had a bilateral orchidectomy minimally three months prior to screening iii. Male participants having a pregnant female partner or a male sexual partner: At least one barrier method has to be used in this case.

   b. Effective contraception methods: i. Female participants: Two methods, including methods that the participant's sexual partner(s) use. At least one must be a barrier method. Contraception must be practised for at least until 12 weeks after the last dose of experimental treatment. For stage 3, female participants of child-bearing potential must have used contraception if any sexual intercourse has occurred after last menses or within the last 3 weeks (whichever is later) before participation, and agree to use non-user dependent contraception: depo-provera injection* or an intrauterine device additional to one barrier method.

   *Including a back-up method of contraception for at least 7 days to prevent unintended pregnancy if injection has been administered within the first 5 days of their menstrual cycle. Otherwise, a back-up barrier method of contraception is required for one month to prevent unintended pregnancy.

   ii. Male participants: Two methods, including methods that the participant's female sexual partner(s) use. At least one must be a barrier method. Effective contraception must be ensured for at least 12 weeks after the last dose of experimental treatment.

   Exclusion Criteria:

<!-- -->

1. Circumstances that raise doubt about free, unconstrained consent to study participation (e.g., person in detention or person with mental disability)
2. Poor general condition where delay in treatment cannot be tolerated or death within four months is likely.
3. Circumstances (in the opinion of the investigator) that raise doubt about ability to complete the follow-up during the study period.
4. The participant is pregnant or breast-feeding or planning to become pregnant in the study period.
5. The participant is infected with HIV with a CD4 count <220 cells/mm3. If >220 cells/mm3, participants will be included only if any of the following is applicable:

   • The participant is antiretroviral (ARV) naïve and able to postpone commencing HIV treatment for 2 months after the trial has started and then restrict regimens to those mentioned in section on ARVs or

   • The participant is ARV experienced (has been on ARV´s a minimum of 5 months), AND: ARV treatment is compliant to, or can be modified as described in the section on Antiretroviral Therapy
6. The participant has a known intolerance to any of the study drugs or concomitant disorders or conditions for which study drugs or standard TB treatment are contraindicated.
7. The participant has a history of, or current evidence of clinically relevant cardiovascular metabolic, gastrointestinal, neurological, hepato-biliary, renal, psychiatric or endocrine diseases, malignancy, or any other condition that will influence treatment response, study adherence or survival in the judgement of the investigator, especially:

   a. Neuropathy, or significant psychiatric disorder like depression or schizophrenia; especially if treatment for those has ever been required or is anticipated to be required b. Evidence of clinically significant extra-pulmonary TB (e.g. miliary TB, TB meningitis, but not limited lymph node involvement) c. Serious lung conditions other than TB, or significant respiratory impairment in the discretion of the investigator d. Uncontrolled diabetes mellitus or diabetes mellitus receiving/requiring treatment with metformin or sulfonylureas e. Cardiovascular disease such as myocardial infarction, heart failure, coronary heart disease, arrhythmia, tachyarrhythmia, or pulmonary hypertension f. Uncontrolled arterial hypertension (systolic blood pressure ≥150 mmHg and/or diastolic blood pressure of ≥95 mmHg on two occasions during screening. An attempt at antihypertensive treatment during the screening period is permitted).

   g. Long QT syndrome or family history of long QT syndrome or family history of sudden death of unknown or cardiac-related cause h. Alcohol, regular opiate, or other drug abuse that is sufficient to significantly compromise the safety or cooperation of the participant, that includes substances prohibited by the protocol or has led to significant organ damage at the discretion of the investigator; AND/OR any abuse of methamphetamine.

   i. History of optic neuropathy j. Vitiligo
8. Any of the following laboratory findings at screening:

   a. Serum amino aspartate transferase (AST) and/or alanine aminotransferase (ALT) >3x the upper limit of normal (ULN), b. Serum alkaline phosphatase or y-glutamyl transferase > 2.5x the ULN, c. Serum total bilirubin level >1.5x the ULN d. Estimated creatinine clearance -eCrCl (using the CKD-EPI 2021 creatinine formula):

   - Stage 1: Lower than 30 ml/min)

   - Stage 2: Lower than 30ml/min or lower than 60 ml/min in participants living with HIV

   - Stage 3: Lower than 80ml/min e. Proteins in urine dipstick >=2+ f. Haemoglobin level <7.0 g/dl g. Platelet count <50,000/mm3, h. Serum potassium below 3 mmol/l, persisting after correction.
9. ECG findings in the screening ECG: (one or more):

   1. QTcF of >450 milliseconds
   2. Atrioventricular (AV) block with PR interval > 200 milliseconds
   3. QRS complex > 120 milliseconds
   4. Any other changes in the ECG that are clinically relevant as per discretion of the investigator
10. Restricted medication:

    1. Treatment with any other investigational drug within 2 month prior to enrolment or enrolment into other clinical (intervention) trials during participation.
    2. Previous anti-TB treatment with drugs active against MTB within the last 3 months prior to screening.
    3. Unable or unwilling to abide by the requirements regarding restricted medication or have taken restricted medication. Restricted medication includes the following drug classes, with relevant timing of intake, and possible exceptions. Exceptions may be permissible after discussion with the sponsor medical expert.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to stable culture conversion to negative in liquid media | Day 01- Week 26
  The primary efficacy endpoint of arms 1 and 2 will be time to stable culture conversion to negative in liquid media defined as the time from enrolment to the first of two negative weekly sputum cultures without an intervening positive culture in liquid media, in comparison to arm 3.
  The efficacy of BTZ-043 will be evaluated by measuring the change in mycobacterial load over time on treatment as quantified by time to positivity in BD MGIT 960® liquid culture described by non-linear mixed-effects methodology, in comparison to arm 3.
Change in Mycobacterial load (Stage 3) | Baseline until week 12 of treatment.
  The efficacy of the arms 5 and 6 (Stage 3) will be evaluated by measuring the change in mycobacterial load over time on treatment as quantified by time to positivity in BD MGIT 960® liquid culture described by non-linear mixed-effects methodology, in comparison to arm 7 using the TTP0-8 or 12 weeks slope.

SECONDARY OUTCOMES:
Relapse - free survival at 12 months after randomization | Day 01-364
  To assess treatment efficacy based on proportion of patients with relapse free outcome at 12 months after randomization.
  Sustained cure at 12 months (52 weeks) after randomization without a failure or relapse event is achieved when all the following criteria are met:
  * known to be alive at or after 48 weeks after randomization;
  * having Sustained Culture Negativity at 48 weeks after randomization;
  * not having met criteria for Failure or Relapse event (see below);
  * not in need of TB treatment and having had no substantial treatment modifications or additional treatment for TB outside of the pre-specified treatment strategies.
Frequency of all adverse events (serious and non-serious) | Day 01-182
  To assess the frequency, severity, and type of adverse events (AEs), and AE related treatment discontinuations.
Frequency of adverse events of Grade 3 severity (severe) or higher | Day 01-182
  Severity of AEs will be classified following the U.S. National Institutes of Health Common Terminology Criteria for Adverse Events 5.0 (CTCAE). The minimum grade is 1 (Mild) and the maximum grade is 5 (Death related to AE). Higher scores mean a worse outcome.
Frequency of adverse events possibly, probably or definitely related to study drug | Day 01-182
  To assess the frequency, severity, and type of adverse events (AEs), and AE related treatment discontinuations.
Frequency of treatment discontinuations or interruptions related to adverse events/serious adverse event | Day 01-182
  To assess the frequency, severity, and type of adverse events (AEs), and AE related treatment discontinuations.
Changes in ECG intervals of PR, RR, QRS, QT, Fridericia-corrected QT [QTcF] | Day 01-182
  * Proportion of participants with QTcF > 500ms in ECGs on treatment
  * Proportion of participants who have a QTcF prolongation of grade 3 or higher
Area under the plasma concentration curve from dosing to the end of the dosing interval (AUC 0-24) predicted from limited pharmacokinetic sampling. | Day 14
  For RIF, PZA, MXF, and IHN (arms 1-3), and BTZ-043, RIF, INH and PZA (arm 4) in all participants with limited pharmacokinetic sampling strategy being done on WK 02 (Day 14 ± 2 Days).
The observed maximum concentration (Cmax) | Day 14
  For RIF, PZA, MXF, and IHN (arms 1-3), and BTZ-043, RIF, INH and PZA (arm 4) in all participants with limited pharmacokinetic sampling strategy being done on WK 02 (Day 14 ± 2 Days).
Time to reach Cmax (Tmax) | Day 14
  For RIF, PZA, MXF, and IHN (arms 1-3), and BTZ-043, RIF, INH and PZA (arm 4) in all participants with limited pharmacokinetic sampling strategy being done on WK 02 (Day 14 ± 2 Days).
Minimum observed plasma concentration 24 hours following the last dose (Cmin) | Day 14.
  For RIF, PZA, MXF, and IHN (arms 1-3), and BTZ-043, RIF, INH and PZA (arm 4) in all participants with limited pharmacokinetic sampling strategy being done on WK 02 (Day 14 ± 2 Days).
DTG and TFD concentration | Day 01-15
  concentrations will be compared at screening and at week 2. More time points may be determined if leftover samples are available. Timing of last DTG and TFD dose intake will be recorded.
Identification of M. tuberculosis complex and Rifampicin (RIF) resistance by PCR (GeneXpert Ultra MTB/RIF®/GeneXpert XDR/HAIN MTBDRplus or similar) | Day 01-182
  Cultures grown from the screening period, and the last sputum sample with mycobacteriological growth will be assessed. This test is qualitative, therefore the result will be: Detected, not detected or indeterminate.
Identification of M. tuberculosis complex and Isoniazid (INH) resistance by PCR (GeneXpert Ultra MTB/RIF®/GeneXpert XDR/HAIN MTBDRplus or similar) | Day 01-182
  Cultures grown from the screening period, and the last sputum sample with mycobacteriological growth will be assessed. This test is qualitative, therefore the result will be: Detected, not detected or indeterminate.
Minimum inhibitory concentrations (MIC) of study drugs the patient was receiving | Day 01-182
  Cultures grown from the screening period, and the last sputum sample with mycobacteriological growth will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hoelscher, Prof Dr., Study Director — LMU University Hospital
Locations (10):
- Centre de Recherches Médicales de Lambaréné (CERMEL), Lambaréné, Gabon
- Kamuzu College of Health Sciences (formerly College of Medicine), Blantyre, Malawi
- Instituto Nacional de Saúde (INS), Maputo, Mozambique
- South Africa (3):
  - Isango Lethemba TB Research Unit. Clinical HIV Research Unit (CHRU), Wits Health Consortium., Port Elizabeth, Eastern Cape
  - TASK Applied Sciences Clinical Research Centre, Cape Town
  - University of Cape Town Lung Institute, Cape Town
- Tanzania (3):
  - National Institute for Medical Research (NIMR-MMRC), Mbeya, Mbeya
  - Ifakara Health Institute (IHI), Bagamoyo
  - Kilimanjaro Clinical Research Institute (KCRI), Moshi
- Makerere University Lung Institute Limited, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No
Currently exploring data sharing via the TB CAPT research data repository.